CLINICAL TRIAL: NCT04500613
Title: Utilization of Erector Spinae Plane Blocks in a Multimodal Analgesic Pathway for Instrumentation and Fusion of Adolescent Idiopathic Scoliosis: A Feasibility Study
Brief Title: Erector Spinae Plane Blocks for Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-2131
Record Dates: First submitted 2020-07-27; First posted 2020-08-05 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative; Opioid Use; Recruitment
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB with Bupivacaine and Dexamethasone (Active Comparator): 12 pediatric spinal fusion surgery patients will be randomized to receive intraoperative ultrasound-guided bilateral ESPB with 0.25% bupivacaine with 2mg preservative free dexamethasone with a maximum of 30 mL total per side, depending on the patient's weight.
  Interventions: Procedure: Bilateral Erector Spinae Plane Block with bupivacaine and dexamethasone
- No ESPB (Placebo Comparator): 12 pediatric spinal fusion surgery patients will be randomized to not receive an intraoperative ultrasound-guided bilateral ESPB. These patients will still receive the standard anesthesia regimen during and after surgery.
  Interventions: Other: No bilateral Erector Spinae Plane Block (no bupivacaine and no dexamethasone)

INTERVENTIONS:
Procedure: Bilateral Erector Spinae Plane Block with bupivacaine and dexamethasone — Bupivacaine is administered typically to reduce sensation in an area. It acts as a nerve block for surgical procedures. Dexamethasone is a corticosteroid that reduces inflammation.
  Arms: ESPB with Bupivacaine and Dexamethasone
Other: No bilateral Erector Spinae Plane Block (no bupivacaine and no dexamethasone) — Patients who are randomized to this group will not receive a bilateral erector spinae plane block
  Arms: No ESPB

SUMMARY:
Pediatric spinal fusion (PSF) surgery is a painful procedure that can treat adolescent idiopathic scoliosis (AIS). One technique that can potentially reduce patients' pain levels and need for opioid medication is the ultrasound-guided Erector Spinae Plane Block (ESPB). The ESP block is a technique that involves injecting an anesthetic medication into the muscles of the lower back on both sides of the spine. Previous studies have shown that ESPB application led to a reduction in opioid use, and there is one pediatric case report of ESPB use in two patients undergoing PSF. However, there is still lack of evidence that the ESPB technique is feasible and effective in the pediatric patient population.

The present study is designed to be the first randomized controlled trial to evaluate the role of ESPB in pediatric spinal fusion surgery and the role of ESPB within an enhanced recovery pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-19 years old
* Patients undergoing multilevel posterior spinal instrumentation and fusion
* Undergoing surgery for correction of adolescent idiopathic scoliosis
* Patients under the care of participating surgeons
* English Speaking

Exclusion Criteria:

* Patients younger than 10 years old or older than 19 years old
* Neuromuscular scoliosis
* Patient under the care of non-participating surgeon performing the procedure
* History of chronic opioid therapy (longer than 4 weeks) to treat back pain attributed to scoliosis tolerance, as defined by Centers for Disease Control (CDC) criteria (more than 60 oral morphine equivalents (OME) daily for over 2 weeks)
* Chronic pain conditions necessitating neuromodulating medications (gabapentin, pregabalin)
* Allergy, intolerance, or contraindication to any protocol component/study medication/technique
* Patient or parent refusal
* Non-english speaking

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Ruby, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery (HSS), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Started | 12 | 12
Completed | 9 | 12
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: One patient was excluded from analysis due to a surgically induced change unrelated to the ESPB, resulting in abortion of surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (2.1) | 15.1 (2.3) | 14.9 (2.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 6 | 7 | 13
  Gender: Male | 4 | 5 | 9
  Gender: Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Receive Bilateral, Pre-incision ESPB
Description: number who receive the intervention and complete all assessments
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 12 | 12
Participants | 9 | 12

2. Secondary Outcome: Rate of Recruitment
Description: Number enrolled and allocated to specific group
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

3. Secondary Outcome: Blinding Assessment
Description: Based on Bang's Blinding Index. Patients' ability to determine whether or not they received the ESPB. The success of patient blinding in each group will be quantified using the Bang Blinding Index which ranges from -1 to 1. Scores closest to 0 indicate a less likelihood that patients were able to guess which group they were randomized into. A score of 1 or -1 means that patients were able to guess which group they were in or guessed the wrong group, respectively. This value is obtained by asking patients which group they believe they were randomly assigned to.
Time Frame: 24 hours after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
score on a scale | 0 [-.30 to .30] | -0.33 [-.63 to -0.04]

4. Secondary Outcome: Number of Participants Unable to Receive ESPB Block.
Description: Number of participants who were randomized to receive the ESPB block, but were unable to receive the block. The no ESPB group were randomized not to get the ESPB block, leading to 0 instances of missed ESPB block.
Time Frame: Holding area, Post-Anesthesia Care Unit (PACU) (hour 0), hour 8, 12, and 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
Participants | 2 | 0

5. Secondary Outcome: Attrition
Description: Number of patients who enroll but do not receive the intervention and/or study assessments.
Time Frame: through study completion, an average of 1 year
Measure: Number; unit: participants
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 12 | 12
participants | 3 | 0

6. Secondary Outcome: Incidence of Intra- and Postoperative Complications Attributed to ESPB
Description: Interference with intraoperative neuromonitoring, infection, local anesthetic toxicity, bleeding/hematoma, extremity weakness
Time Frame: During surgery, PACU (hour 0), hour 8, 12, and 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

7. Secondary Outcome: Pain Scores at Rest and Movement
Description: Measured by Numeric Rating Scale (NRS) pain at rest and with movement (0 being no pain and 10 being as bad as you can imagine). NRS was collected for each participant, Mean and Standard Deviations are found below.
Time Frame: PACU (Post Anesthesia Care Unit, hour 0), hour 8, 12, and 24 hours after surgery, and at hospital discharge (an average of 4 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
score on a scale
  NRS upon PACU Arrival | 3.64 (3.93) | 3.58 (4.19)
  NRS at 8 Hours | 4 (3.37) | 2.5 (1.62)
  NRS at 12 Hours | 3.3 (2.45) | 3 (3.36)
  NRS at rest at 24 hours | 3.55 (1.63) | 2.42 (2.19)
  NRS with Movement at 24 Hours | 5.82 (2.44) | 5 (2.66)
  NRS at rest at Discharge | 3.36 (1.5) | 3 (1.95)
  NRS with movement at Discharge | 4.09 (2.07) | 3.18 (1.66)

8. Secondary Outcome: Total Opioid Consumption
Description: Measured in mean oral morphine equivalents (OME)
Time Frame: 0-24 hours after surgery (OME within 24 hrs)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
milligrams | 78.23 (31.52) | 53.89 (27.68)

9. Secondary Outcome: Time to First Opioid Use
Description: Time to pressing Intravenous Patient-Controlled Analgesia (IV PCA) and to requesting first oral opioid
Time Frame: Up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
minutes | 178 [43 to 309] | 94 [57.5 to 246.5]

10. Secondary Outcome: Opioid Related Side Effects
Description: Measured by 10 symptom Opioid Related Symptom Distress Scale (ORSDS). Frequency of each symptom within the cohort was assessed.
Time Frame: 24 hours after surgery
Measure: Number; unit: participants
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 12
participants
  Fatigue | 3 | 9
  Drowsiness | 6 | 7
  Concentration | 1 | 2
  Nausea | 7 | 10
  Dizziness | 6 | 8
  Constipation | 0 | 1
  Itching | 4 | 2
  Urination | 0 | 0
  Confusion | 1 | 2
  Vomiting | 3 | 5

11. Secondary Outcome: Patient/Parent Satisfaction With Pain Management
Description: Measured via Likert rating scale (0 being strongly dissatisfied and 10 being strongly satisfied)
Time Frame: At hospital discharge (an average of 4 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
Number analyzed (Participants) | 11 | 10
score on a scale
  Patient | 10 [7 to 10] | 8 [7 to 10]
  Parent | 10 [9 to 10] | 9 [8 to 10]

ADVERSE EVENTS:
Time Frame: Throughout the completion of the study, approximately 1 year
Arm/Group | ESPB With Bupivacaine and Dexamethasone | No ESPB
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04500613/Prot_SAP_000.pdf